CLINICAL TRIAL: NCT06398509
Title: Futuros Fuertes 2.0 A Primary Care Based Intervention to Prevent Obesity Among Low-income Latino Children
Brief Title: A Primary Care Based Intervention to Prevent Childhood Obesity Among Low-income Latino Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-38707; 1R01HD109158 (NIH)
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Futuros Fuertes 2.0 intervention includes brief health education and coaching at well child visits in the first two years of life that addresses optimal feeding, screen time and sleep practices. In addition, caregivers receive 2 text messages per week. Caregivers also receive environmental prompts to help support healthy behaviors at home.
  Interventions: Behavioral: Futuros Fuertes 2.0
- Control (Active Comparator): The control intervention includes brief health education and coaching at well child visits in the first two years of life that addresses home safety, management of common childhood illnesses, and promotion of language development. In addition, caregivers receive 2 text messages per week. Caregivers also receive environmental prompts to help support healthy behaviors at home.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Control — The control intervention includes brief health education and coaching sessions just after well child visits in the first two years of life (total of 7 sessions), 2 text messages per week for the primary caregiver and up to two additional family members, and environmental prompts that support healthy behaviors. The control intervention focuses on home safety, home management of common childhood illnesses, and promotion of language development.
  Arms: Control
Behavioral: Futuros Fuertes 2.0 — The Futuros Fuertes 2.0 intervention includes brief health education and coaching sessions just after well child visits in the first two years of life (total of 7 sessions), 2 text messages per week for the primary caregiver and up to two additional family members, and environmental prompts that support healthy behaviors. The Futuros Fuertes 2.0 intervention focuses on optimal infant feeding, screen time, and sleep practices.
  Arms: Intervention

SUMMARY:
The goal of this study is to evaluate the impact of a primary care based intervention to promote optimal feeding, screen time and sleep practices among low-income Latino infants and toddlers. Infants and caregivers will receive brief health education and coaching sessions from health educators at primary care visits in the first two years of life as well as two text messages per week with health information and tips. Half of the participants will receive the Futuros Fuertes 2.0 intervention that includes health coaching and education on infant feeding, screen time and sleep (intervention group). The other half will receive health coaching and education on safety, home management of childhood illnesses, and promotion of language development (control group). We will look at the impact of the Futuros Fuertes 2.0 intervention on child BMI and various health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Parent/caregiver self identifies as Latino
* Parent/caregiver speaks Spanish or English
* Parent/caregiver intends to receive primary care for infant at participating clinic
* Infant gestational age of 37 weeks or greater
* Infant birthweight of 2600 grams or greater
* For multiples (twins, triplets), one sibling will be chosen at random to participate

Exclusion Criteria:

-Infant has a serious medical condition that affects feeding or growth

Ages: 7 Days to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 576 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
BMI Z-score | 24-months
  BMI Z-score based on WHO growth curves

SECONDARY OUTCOMES:
Breastfeeding | First year of life
  Duration of breastfeeding in first year of life
Screen time | 24-months
  Daily screen time
Sleep duration | 24-months
  Daily sleep duration
Fruit and vegetable intake | 24-months
  Daily fruit and vegetable intake
Sugar sweetened beverage and 100% fruit juice intake | 24-months
  Weekly ounces of sugar-sweetened beverages and 100% fruit juice
Change in BMI Z-score | 6-months to 24-months
  Trajectory of BMI Z-score (WHO growth curve)

OTHER OUTCOMES:
Screen time | 6-months, 12-months and 18-months
  Daily screen time
Sleep duration | 6-months, 12-months, 18-months
  Daily sleep duration
Sugar-sweetened beverages and 100% fruit juice | 6-months, 12-months, 18-months
  Weekly ounces of sugar-sweetened beverages and 100% fruit juice

CONTACTS AND LOCATIONS:
Overall Officials: Amy Beck, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Children's Health Center San Francisco General Hospital, San Francisco, California
  - Valley Health Center Sunnyvale, Sunnyvale, California

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, final research data will be available for use by other investigators, federal agencies, or other appropriate organizations or personnel upon request. Research data will be shared in a de-identified data set to protect subject privacy.